CLINICAL TRIAL: NCT04061928
Title: The Combination of Toripalimab With Preoperative Chemoradiotherapy for Locally Advanced Adenocarcinoma of Esophagogastric Junction
Brief Title: Toripalimab With Preoperative Chemoradiotherapy for LA-EGJ
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Ziyu Li, MD, The director of ward 1 of gastrointestinal tumor center, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019YJZ38
Record Dates: First submitted 2019-08-01; First posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: PD-1; Chemoradiotherapy; Gastroesophageal Junction Cancer
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of toripalimab with preoperative chemoradiotherapy (Experimental): This is a one arm study, enrolled locally advanced EGJ patients will receive toripalimab and combined with preoperative chemoradiotherapy and operation.
  generic name：PD-1 dosage form：Injection dosage：240mg (6ml) frequency：every 3 weeks duration：4 times before operation and 4 times after operation
  Interventions: Drug: PD-1

INTERVENTIONS:
Drug: PD-1 — 2 times PD-1 (240mg) combined with preoperative chemoradiotherapy，then another 2 times PD-1 before operation. 4 times PD-1 combined with postoperative chemotherapy.
  Other Names: Toripalimab

SUMMARY:
This study aims to investigate the safety and efficacy of radiotherapy combined with Toripalimab (PD-1 inhibitor) in the treatment of locally advanced adenocarcinoma of the gastroesophageal junction.

DETAILED DESCRIPTION:
In this study, patients with locally advanced adenocarcinoma of gastroesophageal junction will be enrolled to explore the safety and efficacy of preoperative radiotherapy and chemotherapy combined with Toripalimab (PD-1). Around 45 patients will be recruited in this one-arm cohort. All patients in this cohort will be treated with preoperative radiotherapy and chemotherapy plus PD-1 for two times, then another two times of PD-1 before operation. After surgery, postoperative chemotherapy plus PD-1 will be carried out for four times. This study focuses on the safety of chemoradiotherapy combined with immunotherapy, and whether the TRG grade, LC, DFS have been improved.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 18-75, male and female.

  2) ECOG score was 0-1.

  3) Diagnosis of adenocarcinoma in the gastroesophageal junction.

  4) Initial treatment of locally advanced patients (cT3-4 or N+, and M0).

  5) The estimated survival time will be more than 12 months.

  6) Adequate organ reserve function.

  7) agree to join the group, willing to cooperate with clinical research, and sign the informed consent.

Exclusion Criteria:

* 1) Patients have received immunotherapy, such as PD-1 antibody, PD-L1 antibody and CTLA4 antibody.

  2) Immunosuppressive drugs were used within 4 weeks before admission.

  3) Active infection, acute myocardial infarction in recent 6 months, severe arrhythmia requiring long-term drug intervention, severe stroke, uncontrolled epilepsy or other serious medical complications.

  4) In the past five years, there have been other malignant diseases except for cured skin cancer and cervical cancer in situ.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-08-26 (Estimated); Primary Completion 2022-08-25 (Estimated); Study Completion 2023-08-25 (Estimated)

PRIMARY OUTCOMES:
TRG (Tumor Regression Grading) | 10 days after operation
  The TRG of operation after neoadjuvant chemoradiotherapy and immunotherapy.

SECONDARY OUTCOMES:
Number of participants with AEs (Adverse Events) | Through study completion, an average of 1 year
  The AEs during the trial, including radiation mucositis, bone marrow suppression, AEs related to immunotherapy and so on
LC (Local Control) | Through study completion, an average of 1 year
  The local control of the patients
DFS (Disease Free Survival) | Through study completion, an average of 1 year
  The disease free survival of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Ziyu Li, MD, Principal Investigator — Peking University Cancer Hospital & Institute; Yongheng Li, MD, Principal Investigator — Peking University Cancer Hospital & Institute

IPD SHARING:
Plan to Share IPD: No